CLINICAL TRIAL: NCT06501638
Title: Efficacy and Safety of memanTine in the Treatment Of Frequently symPtomatic Atrial Premature Beats: a Multicenter Randomized Double-blind Placebo-controlled Study
Brief Title: Efficacy and Safety of memanTine in the Treatment Of Frequently symPtomatic Atrial Premature Beats
Acronym: STOP-AP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Yihan Chen, Professor, Shanghai East Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024YS-146
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Atrial Premature Beats, Contractions, or Systoles
Keywords: Atrial Premature Beats; memantine; double-blinded; randomized; placebo control
MeSH Terms: conditions — Atrial Premature Complexes | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memantine (Experimental): Take Memantine Hydrochloride for intervention
  Interventions: Drug: Memantine Hydrochloride 10 MG
- Placebo (Placebo Comparator): Take placebo for intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine Hydrochloride 10 MG — Take Memantine Hydrochloride for intervention First week, 5mg(half the tablet), p.o.，bid. Second to Sixth week, 10mg(one tablet), p.o., bid
  Arms: Memantine
Drug: Placebo — Take placebo for intervention First week, half the tablet, p.o., bid. Second to Sixth week, one tablet, p.o., bid
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled study to expIore the efficacy and safety of Memantine hydrochIoride tabIets to treat patients with frequent PACs.

DETAILED DESCRIPTION:
After preliminary screening, the target patients will undergo continuous 3-day (72-hour) monitoring with a wearable holter patch(as baseline data) to assess the number of baseline atrial premature beats. Based on the monitored data, it will be determined whether the subjects meet the inclusion criteria. Eligible participants will be randomly assigned in a 1:1 ratio (on Day 0) to either the experimental group (administered with hydrochloride memantine tablets) or the control group (placebo). A total of 256 subjects will be enrolled, with 128 subjects in each group, stratified by age (age ≥ 65 years vs. age < 65 years) and the number of atrial premature beats (≥ 5000 beats/24h vs. < 5000 beats/24h).

The subjects in the experimental group will take hydrochloride memantine tablets according to the following regimen:Week 1: Half tablet per dose (5mg/dose), twice daily, taken orally at the same time in the morning and evening (with a recommended dosing interval of 12 hours ± 2 hours).Week 2 to Week 6: One tablet per dose (10mg/dose), twice daily, taken orally at the same time in the morning and evening (with a recommended dosing interval of 12 hours ± 2 hours).

Control group (placebo): The subjects in the control group will take placebo according to the following regimen:Week 1: Half tablet per dose, twice daily, taken orally at the same time in the morning and evening (with a recommended dosing interval of 12 hours ± 2 hours).Week 2 to Week 6: One tablet per dose, twice daily, taken orally at the same time in the morning and evening (with a recommended dosing interval of 12 hours ± 2 hours).

The study consists of a screening period (D0-D7 days), a treatment period (D8-D42 days), and a follow-up period (D43-D56 days).The start dates for the 3-day ambulatory holter patch are as follows: D25-D28, D39-D42, and D53-D56.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 (inclusive).
2. Presence of symptoms related to premature atrial contractions (PACs) during screening, with PACs occurring ≥1000 times/24 hours.
3. Understanding and willingness to comply with the study procedures and methods, voluntary participation in the study, and signing an informed consent form.

Exclusion Criteria:

1. Atrial fibrillation, atrial flutter, or persistent atrial tachycardia (confirmed by electrocardiogram within the past 6 months or detected by continuous 3-day (72h) monitoring with a wearable Holter monitor at baseline); or ventricular tachycardia (excluding occasional short episodes of ventricular tachycardia during sleep) or ventricular fibrillation.
2. Occurrence of a stroke event, including hemorrhagic/ischemic stroke and transient ischemic attack (TIA), within the past 6 months prior to screening; history of cardiac surgery, myocardial infarction (MI), percutaneous coronary intervention (PCI), or atrial arrhythmia radiofrequency ablation within the past 3 months prior to screening.
3. Left ventricular ejection fraction (LVEF) ≤40%; or New York Heart Association (NYHA) functional class III or IV.
4. Sick sinus syndrome, second-degree type II or higher atrioventricular block, or bifascicular block without permanent pacemaker implantation.
5. Ongoing use of amiodarone within the past 4 weeks prior to screening, or ongoing use of antiarrhythmic drugs other than amiodarone, as well as Chinese herbal medicine with antiarrhythmic effects within the past 1 weeks prior to screening.
6. Presence of unstable angina, severe congenital heart disease (excluding patent foramen ovale), post-artificial heart valve replacement, acute myocarditis, acute endocarditis, rheumatic heart valve disease,Hypertrophic obstructive cardiomyopathy.
7. Coexistence of other diseases with an expected survival period of less than 1 year.
8. Active hepatitis or significant liver dysfunction (ALT or AST >3 times the upper limit of normal [ULN], TBIL >3 ULN).
9. Severe renal insufficiency (calculated estimated glomerular filtration rate [eGFR] <40 ml/min/1.73m² using the CKD-EPI equation).
10. Received investigational drugs or medical device treatments in other clinical trials within 1 month prior to screening or within 5 half-lives (whichever is longer).
11. Pregnancy, lactating women, or positive pregnancy test result before randomization.
12. Hyperthyroidism that has not been properly treated and thyroid function has not returned to normal, the perioperative period of cardiothoracic surgery (one week before surgery to two weeks after surgery), uncorrected electrolyte disturbances (serum K+ > 5.5 mmol/L or < 3.5 mmol/L, serum magnesium < 1.5 mmol/L, etc.); chronic obstructive pulmonary disease (COPD) combined with respiratory failure or infection that has not been corrected, etc.
13. History of epilepsy, seizures, or mental illness.
14. Known allergy to memantine hydrochloride tablets or their excipients.
15. Patients currently receiving memantine treatment for moderate or severe Alzheimer's disease.
16. Other circumstances where the investigator deems the subject unsuitable for inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
percentage reduction of 24-hour premature atrial beats count | The sixth week after intervention
  Participants accepted 3-day holter patch monitor at baseline, fourth, sixth and eighth week after intervention. Average 24-hour premature atrial beats count was then calculated.
  percentage reduction of 24-hour premature atrial beats count = (24-hour premature atrial beats count(baseline)-24-hour premature atrial beats count (sixth week) ) /24-hour premature atrial beats count(baseline)

SECONDARY OUTCOMES:
change of 24-hour premature atrial beats count | The fourth, sixth and eighth week after intervention
  Participants accepted 3-day holter patch monitor at baseline, fourth, sixth and eighth week after intervention. Average 24-hour premature atrial beats count was then calculated.
  change of 24-hour premature atrial beats count =24-hour premature atrial beats count(baseline)-24-hour premature atrial beats count (observation time)
change of 24-hour premature atrial beats burden | The fourth, sixth and eighth week after intervention
  Participants accepted 3-day holter patch monitor at baseline, fourth, sixth and eighth week after intervention. Average 24-hour premature atrial beats burden was then calculated.
  change of 24-hour premature atrial beats burden =24-hour premature atrial beats burden(baseline)-24-hour premature atrial beats burden (observation time)
change of 24-hour non-sustained atrial tachycardia episodes | The fourth, sixth and eighth week after intervention
  Participants accepted 3-day holter patch monitor at baseline, fourth, sixth and eighth week after intervention. Average 24-hour premature atrial beats episodes was then calculated.
  change of 24-hour non-sustained atrial tachycardia episodes=24-hour non-sustained atrial tachycardia episodes (baseline)- 24-hour non-sustained atrial tachycardia episodes (observation time)
change of 24-hour non-sustained atrial tachycardia burden | The fourth, sixth and eighth week after intervention
  Participants accepted 3-day holter patch monitor at baseline, fourth, sixth and eighth week after intervention. Average 24-hour non-sustained atrial tachycardia burden was then calculated.
  change of 24-hour non-sustained atrial tachycardia burden =24-hour non-sustained atrial tachycardia burden(baseline)- 24-hour non-sustained atrial tachycardia burden (observation time)
change of 24-hour sustained atrial tachycardia, atrial flutter and atrial fibrillation episodes | The fourth, sixth and eighth week after intervention
  Participants accepted 3-day holter patch monitor at baseline, fourth, sixth and eighth week after intervention. Average 24-hour sustained atrial tachycardia, atrial flutter and atrial fibrillation episodes was then calculated.
  change of 24-hour non-sustained atrial tachycardia episodes=newly discovered 24-hour non-sustained atrial tachycardia episodes (observation time)
The proportion of new-onset persistent atrial tachycardia, atrial fibrillation (AF), and atrial flutter during continuous 72-hour monitoring at weeks 4, 6, and 8 | The fourth, sixth and eighth week after intervention
  The proportion of subjects with persistent atrial tachycardia, AF, and atrial flutter ≥ 30 seconds first recorded during the planned continuous 72-hour electrocardiographic monitoring at weeks 4, 6, and 8.This endpoint will be calculated based on the first occurrence of SAT, AF, or AFL during the respective 72-hour monitoring windows;
Cumulative incidence of new-onset AF from week 0 to week 8: | The eighth week after intervention
  the proportion of subjects with AF ≥ 30 seconds first recorded at any follow-up window at weeks 4, 6, and 8 from randomization to the end of week 8. If the same subject has AF at weeks 4, 6, the first occurrence of AF is counted as one case, with a maximum of one count per subject
SF-36 score change | The sixth week after intervention
  Participants accepted the Mos 36-item Short Form Health Survey evaluation at baseline and sixth after intervention.
  SF-36 score change= SF-36 score (baseline)-SF-36 score (sixth week)
Efficacy analysis of atrial premature beats or non-sustained atrial tachycardia | The fourth, sixth and eighth week after intervention
  Efficacy Criteria for Atrial Premature Beats Treatment:
  A reduction of ≥50% in the average number of atrial premature beats over 24 hours compared to baseline after taking the study drug (Memantine Hydrochloride Tablets or placebo).
  Efficacy Criteria for Non-sustained Atrial Tachycardia Treatment:
  A reduction of ≥50% in the average burden of non-sustained atrial tachycardia over 24 hours compared to baseline after taking the study drug (Memantine Hydrochloride Tablets or placebo).
Safety profile of memantine in patients with frequent symptomatic PACs | The eighth week after intervention
  The incidence of adverse events (including psychiatric symptoms, seizures, bradycardia, new-onset heart failure, etc.), serious adverse events, laboratory test abnormalities, and abnormal electrocardiogram findings.

CONTACTS AND LOCATIONS:
Overall Officials: Yihan Chen, Doctor, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (5):
  • Study Protocol: V2.2 (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT06501638/Prot_001.pdf
  • Study Protocol: V2.3 (2025-06-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT06501638/Prot_002.pdf
  • Study Protocol: V2.1 (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT06501638/Prot_000.pdf
  • Statistical Analysis Plan: V2.0 (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT06501638/SAP_004.pdf
  • Statistical Analysis Plan: V1.0 (2025-02-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT06501638/SAP_003.pdf